CLINICAL TRIAL: NCT04909567
Title: Optimization of Patients' Physical and Mental Status Prior to Colorectal Cancer Surgery -a Randomized Clinical Trial
Brief Title: Optimization of Patients' Physical and Mental Status Prior to Colorectal Cancer Surgery
Acronym: OPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ulf Oskar Gustafsson, MD, PhD, Associate Professor of Surgery, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RCT: OPTIMIZATION: 2021:9
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Complication,Postoperative; ERAS
Keywords: ERAS; RCT; Optimisation
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Optimisation:
  Diet, organised exercise, psychosocial support
  Interventions: Behavioral: Optimisation
- Control arm (No Intervention): Current standard preparation before surgery

INTERVENTIONS:
Behavioral: Optimisation — Defined optimisation
  Arms: Intervention arm

SUMMARY:
Colorectal cancer is one of the most common cancers globally. A majority are operated on for the purpose of cure. Complications after surgery are common, involve long length of stay and increase the risk of later recurrence of cancer. Optimization of physical and mental function before surgery can reduce the risk of complications and provide a faster recovery. However, a standardized form for how optimization should be performed does not exist.

At Danderyd Hospital, Stockholm, Sweden, we are starting up an optimization center where patients are offered optimizing measures while waiting for surgery. This form of structured treatment has not been studied before and we therefore want to investigate outcomes in a randomized study.

All patients with colorectal cancer who are being examined for surgery are offered participation in the study. Randomization of 518 patients in to either an intervention group where the patients; are optimized for concomitant diseases, treated for malnutrition and overconsumption of alcohol and tobacco, undergoes an exercise program and receives psychosocial support before surgery, or a control group where patients are prepared for surgery according to current routines. Primary outcome is the difference in severe complications between the groups. Secondary outcome is difference in length of stay as well as fitness and mental well-being before and 30 days after the operation.If optimization before surgery reduces complications and shortens length of stay, the model can also be used by other operating specialties. This may result in a great improvement for the healthcare in general.

DETAILED DESCRIPTION:
A randomized controlled, unblinded study with block stratification for surgical procedures.

Intervention arm:

All patients in the intervention group will be treated in an "optimization center" which constitutes its own physical location at the hospital and functions as a day care unit staffed with doctors, contact nurses, physiotherapists, ERAS nurses and dietitians. An expert team of cardiologists, physiologists, renal physicians and endocrinologists are attached to the unit.

Day 1. (2-12 weeks before the operation). Multipel testing: Clinical status, ASA score, NSQIP score. Alcohol and Smoke score tests. Nutritional score. 6 minute walk test. Psychiatric score tests. If mortality risk >5% according to NSQIP, low performance on walk test, chair stand test. ASA 3-4, HbA1c >50 for non diabetics, >60 for diabetics or (GFR <45) = special attention from the expert team.

Day 2 until one week before surgery:

Home exercise 5 days / week. Organised (physiotherapist) exercise 2 days / week. Dietprogram with close follow-up. Psychosocial support. Smoking and alcohol cessation program

The week before surgery: The same tests as day 1. 30 days posted: The same tests as day 1.

Controlarm: The same tests as for the intervention group, day 1, the week before surgery and 30 days post. No interventions during the period.

The international ERAS database will be used to record data in the study. Consecutive registration of over 300 perioperative variables on each individual patient.

Examples of these variables are basic patient characteristics, preoperative variables such as information before surgery, laxation, nutrition, fluid intake, anemia and glucose optimization. Intraoperative variables such as body temperature, fluid supply, anesthesia method, bleeding, operation time and gastric tube. Postoperative variables such as catheter removal, nutrition, mobilization, nausea, paralytic ileus, specified complications, reoperations and length of stay after surgery. Compliance with the ERAS protocol will be registered.

ELIGIBILITY:
Inclusion Criteria:

* All patients, 18 years or older, with strong suspicion of colorectal cancer

Exclusion Criteria:

* Patients with dementia with severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Serious complications | 30 days
  Can preoperative optimization change the proportion of serious complications after surgery (defined according to Clavien 3b-5) in intervention vs. control arm.
  ) in intervention vs. control arm

SECONDARY OUTCOMES:
Reoperations | 30 days
  Change of proportion of reoperations in intervention vs. control arm
Length of stay (LOS) | 30 days
  Change of LOS (days) in intervention vs. control arm
Working capacity | 2-12 weeks
  Change of walking distance (meter) in intervention vs. control arm (6 minute walk test)
Weight loss | 2-12 weeks
  Change of weight loss (kg) in intervention vs. control arm
Psychosocial status | 2-12 weeks
  Change of points in Hospital and Anxiety scale (HAD) in intervention vs. control arm

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Gustafsson, MD, PhD, Principal Investigator — Karolinska Institutet; Josefin Karlsson, Nurse, Study Chair — Karolinska Institutet
Locations (1):
- Ulf Oskar Gustafsson, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Data Availability Statement
  Due to Swedish legal restrictions and the current ethical approval for the study, data is not publicly available to share, but the research group can provide descriptive data in table form.